CLINICAL TRIAL: NCT03936621
Title: A Phase II Randomized Cross-over Study of the Efficacy and Safety of Omega 3 Fatty Acid Supplements on Lung Cancer-Promoting Inflammatory Markers in Heavy Smokers
Brief Title: Efficacy and Safety of Omega 3 Fatty Acid Supplements on Heavy Smokers
Acronym: Omega
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: H19-00221
Record Dates: First submitted 2019-04-24; First posted 2019-05-03 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Lung Cancer
Keywords: Omega 3; CRP
MeSH Terms: conditions — Lung Neoplasms | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: participants are randomized into 2 study groups. Group 1 Omega 3 fatty acids for 6 months and then off omega 3 fatty acids for the next 6 months. Group 2. No Omega 3 fatty acids for the first 6 months followed by Omega 3 fatty acids for the next 6 months.
Who Masked: Participant
Masking Description: A computer will be used to select participants for each of the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Omega 3 Fatty Acid (Active Comparator): Omega 3 fatty acids for 6 months and then off omega 3 fatty acids for the next 6 months. In the first 6 months, you will be asked to take one capsule of Omega 3 fatty acids with breakfast and 1 with dinner/day for the first week, 2 capsules in the morning and one capsule in the evening for the second week and then 2 capsules with breakfast and 2 with dinner/day for the remaining 24 weeks. In the next 6 months (Months 7 to 12), you will have a blood test for markers of inflammation at the end of Month 7 and at Month 9 and 12 to determine if the anti-inflammatory effects of Omega 3 acids are still there after you have stopped taking it.
  Interventions: Drug: Omega 3 fatty acid
- Group 2: Control Arm (Placebo Comparator): No Omega 3 fatty acids for the first 6 months followed by Omega 3 fatty acids for the next 6 months. You will be asked to have a blood test for markers of inflammation at Month 1, 3 and 6 for markers of inflammation to determine the natural variation of the levels of these markers without Omega 3 fatty acid supplements. In Month 7, you will be asked to take one capsule of Omega 3 with breakfast and 1 with dinner/day for the first week, 2 capsules in the morning and one capsule in the evening for the second week and then 2 capsules with breakfast and 2 with dinner/day for the remaining 24 weeks.
  Interventions: Drug: Omega 3 fatty acid

INTERVENTIONS:
Drug: Omega 3 fatty acid — To evaluate the efficacy of 3.6 g omega 3 fatty acid supplements (2.4 g EPA + 1.2 g DHA)/day for 6 months versus no treatment at reducing the level of C-reactive protein (CRP) in ever smokers at high risk of lung cancer. The primary endpoint of the study is reduction of CRP.
  Other Names: EPA; DHA; Omega 3

SUMMARY:
The study duration is 12 months. The initial enrollment visit will take approximately one hour. The Month 1, 3, 6, 7, 9 and 12 visits will take approximately 30 minutes each. The three telephone visits will take approximately 10 minutes each. The total time commitment to the study will be approximately four and a half hours.

DETAILED DESCRIPTION:
The table below explains what will be done at each study visit:

Prior to Pre-Registration Informed Consent. Questionnaire (asking about your risks for lung cancer, diet and medications including food supplement). Blood test for CRP level

Prior to Registration/Randomization Blood test for CRP level (about 6 ml or 1 teaspoon) Pregnancy test (either blood or urine, for woman with childbearing potential only)

Registration/Randomization Medical history Physical exam (Vital signs/Body height and weight) Receive 3 month supply of Omega 3 fatty acids for treatment first group. Blood tests for Fasting Blood insulin, etc (about 15 ml or 3 teaspoons) Receive a diary to record the amount of study medication you take each day and any side effects you may experience

Week 2 telephone interview Ask about side effects you may be having Ask about other medications you may be taking Review study agent diary

Month 1 visit (you will not be able to eat anything for 10 hours before the appointment) Blood test for Fasting Blood insulin, etc (15 ml or 3 teaspoons) -( All participants)

Treatment Group:

Ask about side effects you may be having Ask about other medications you may be taking Review study medication diary

Month 2, 4, and 5 telephone interview Review diary Ask about side effects you may be having Ask about other medications you may be taking

Month 3 visit (you will not be able to eat anything for 10 hours before the appointment) Physical exam with vital signs Repeat blood tests (about 15 ml or 3 teaspoons) (All participants)

Treatment Group:

Collect unused omega 3 (for treatment group) Receive next 3 month supply of omega 3 (for treatment group) Review study medication diary Ask about side effects you may be experiencing Ask about other medications you may be taking

Month 6 or end of study visit (if left study early for any reason) Physical exam with vital signs Blood tests (about 15 ml or 3 teaspoons) - All participants

Treatment Group:

Review and collect study agent diary Ask about side effects you may be having Ask about other medications you may be taking

Month 7-12 Cross over study Treatment group will become observation group Observation group will become treatment group with the same procedures in month 1 to 6

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 55 and 80 years
* Are a current or former smoker with a 30 pack-year (e.g. one pack of cigarettes a day for 30 years) smoking history or
* Have a greater than 1.51% chance of developing lung cancer in the next six years based on the investigator's risk prediction tool
* Have elevation of a marker of inflammation called C-Reactive Protein (CRP)
* Are capable of providing informed consent to participate in the study

Exclusion Criteria:

* Have been previously diagnosed with lung cancer
* Have had other non-curatively treated cancer outside the lung.
* Have any medical condition, such as severe heart disease (e.g. unstable angina, chronic congestive heart failure), acute or chronic respiratory failure, home oxygen therapy, bleeding disorder, that in the opinion of the investigator could jeopardize your safety during participation in the study or unlikely to benefit from screening due to shortened life-expectancy from the co-existing illnesses
* Are currently taking omega 3 fatty acid supplements

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in CRP levels in participants from both arms | 1 year
  Blood will be collected over the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam, MD, Principal Investigator — BC Cancer Research Ctr

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Derived] Elisia I, Yeung M, Kowalski S, Wong J, Rafiei H, Dyer RA, Atkar-Khattra S, Lam S, Krystal G. Omega 3 supplementation reduces C-reactive protein, prostaglandin E2 and the granulocyte/lymphocyte ratio in heavy smokers: An open-label randomized crossover trial. Front Nutr. 2022 Dec 1;9:1051418. doi: 10.3389/fnut.2022.1051418. eCollection 2022. PMID 36532545